CLINICAL TRIAL: NCT04743531
Title: Bridging Home and Preschool Environments to Promote Healthy Eating and Activity Behaviors and Prevent Obesity in Early Childhood
Brief Title: Healthy Environments Study (HEROs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Colorado, Denver (Other); New Mexico State University (Other); Pennington Biomedical Research Center (Other); Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USDA 2015-68001-23240
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2020-11

CONDITIONS: Health Behavior; Childhood Obesity
Keywords: Early Childhood; Mindful Parenting; Family Intervention; Picky Eating; Motor Development; Diet Quality; Physical Activity
MeSH Terms: conditions — Health Behavior; Pediatric Obesity; Food Fussiness; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Families living in rural Colorado will participate in the HEROs intervention in Fall 2019.
  Interventions: Behavioral: HEROs
- Staggered Intervention (Experimental): Families in the staggered intervention arm will serve as controls for the first intervention arm during Fall 2019. Families the staggered intervention arm will then participate in the HEROs intervention in Spring 2020.
  Interventions: Behavioral: HEROs

INTERVENTIONS:
Behavioral: HEROs — Intervention Description: The intervention will consist of a 6-week family workshop series, held one evening per week for six consecutive weeks. The intervention modules will be delivered by trained researchers at two preschool sites in rural Colorado in Fall 2019 and Spring 2020. The primary caregiver and preschool child will be the targets of the study. Each of the workshops will be structured to include joint caregiver-child activities and programming that is tailored for caregivers and children individually. Caregivers will learn about and engage in activities related to healthy eating and picky eating; physical activity and motor development; and parenting strategies. Children will participate in activities focused on healthful eating and physical activity that supports content their parents are learning.

SUMMARY:
Obesity is a multi-dimensional problem that has roots in infancy and tracks into adulthood. Obesity is represented disproportionately among children and families from low socioeconomic and minority backgrounds, particularly in rural areas that have limited access to food, activity, and health-related services. There is a need for culturally-tailored, effective interventions that can positively impact the environments (home, preschool, community) in which young children grow and develop their eating and activity behaviors. Developing family interventions, particularly for families with limited resources, requires improving caregivers' health literacy and home food/activity environments, and also requires tailoring to accommodate the realities of stressful and unpredictable family settings. The overall objective of this proposed HEROs Study (HEalthy EnviROnments Study) is to develop a companion, technology-based, interactive family intervention that will promote healthy lifestyles for young children in both Head Start and family settings.

DETAILED DESCRIPTION:
This intervention study will test the impact of the intervention through a quasi-experimental staggered implementation pilot design. The aims will test whether the implementation of a parent-child interaction intervention, focusing on eating and activity behaviors, will improve children's eating behaviors, motor performance and parent-child interactions in these domains. This project seeks to answer the following research questions:

1. Do children participating in the family-based intervention demonstrate enhanced PA and eating behaviors?

   * Hypothesis 1.1: Children receiving the family-based intervention will have higher PA levels and enhanced motor skills compared to children in the control group.
   * Hypothesis 1.2: Children receiving the family-based intervention will demonstrate enhanced eating behaviors compared to children in the control group.
2. Can the home environment be improved by parents' self-monitoring of food availability and electronic devices; and the application of mindful parenting strategies?

   * Hypothesis 2.1: Evaluation of food items in the home and electronic devices in the child's bedroom will demonstrate a more positive home environment of participants receiving the family-based HEROs intervention.
   * Hypothesis 2.2: Parents will report more positive parent-child interactions after receiving the family-based HEROs intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults who identify as the primary caregiver of a child enrolled in a Head Start or preschool center ;
* Caregivers who report their child is without disability, illness, or disorder that would significantly affect dietary or activity behaviors (e.g., diabetes, cerebral palsy);
* Participants who communicate in either English or Spanish language.

Exclusion Criteria:

* Caregivers with children who have a disability, illness, or disorder that would significantly affect dietary or activity behaviors.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Change in children's diet behaviors | Baseline (pre-intervention), Month 2 (post-intervention), Month 4 (follow up)
  The Healthy Kids (HK) survey (Townsend et al 2018) examines 23 behaviors in the child's family environment to identify nutrition, activity, and child feeding factors associated with pediatric obesity in low-income populations. Survey responses will be coded using 4 response options per item (4=most healthful; 1=least healthful). Items will be summed into 6 subscales: vegetables, sweetened beverages, activity (screen and physical activity), snacking, energy density, and BMI.
Change in children's gross motor skill scores | Baseline (pre-intervention), Month 2 (post-intervention), Month 4 (follow up)
  The Test of Gross Motor Development-2 (TGMD-2) will be used to assess child's motor skill competence. The TGMD-2 assesses 12 skills: run, gallop, hop, leap, horizontal jump, slide (locomotor skills); and striking a stationary ball, stationary dribble, kick, catch, overhand throw, and underhand roll (object control skills). A research team member will demonstrate the proficient technique to the child, then the child will be asked to perform the skill twice. Researchers will score each attempt to perform the skill based on set criteria (Logan et al 2011).
Change in children's physical activity levels | Baseline (pre-intervention), Month 2 (post-intervention), Month 4 (follow up)
  Children's physical activity levels will be assessed using the cumulative time in sedentary and moderate and vigorous physical activity (MVPA). Data will be collected using the ActiGraph GT9X accelerometer, which participants will be asked to wear for 7 days during each data collection period (baseline, follow up at month 2, follow up at month 4). Sedentary and MVPA cut points for children will be used to measure of the mean amplitude deviation of acceleration [Vaha-Ypya 2015].
Change in children's willingness to try new foods | Baseline (pre-intervention), Month 2 (post-intervention), Month 4 (follow up)
  Children's willingness to try new foods will be conducted using a Tasting Panel, a food preference assessment, with each child. The child will be asked to taste 8 foods in a self-selected order. This panel includes sweet and savory foods, fruits, vegetables, and protein. After tasting a food, children will be asked to place the food in front of one of 3 cartoon faces that best describes how they think the food tasted: a smiling face (yummy), a neutral face (just ok), or a frowning face (yucky). Refusals to taste a food will be recorded [Johnson et al 2019].

SECONDARY OUTCOMES:
Change in child BMI | Baseline (pre-intervention), Month 2 (post-intervention), Month 4 (follow up)
  Children's weight (measured on a digital scale) and height (measured using a portable stadiometer) will be used to determine a BMI using the CDC standardized growth curves.
Change in caregivers' physical activity levels | Baseline (pre-intervention), Month 2 (post-intervention), Month 4 (follow up)
  Caregivers' physical activity levels will be assessed using the cumulative time in sedentary and moderate and vigorous physical activity. Data will be collected using the ActiGraph GT9X accelerometer, which participants will be asked to wear for 7 days during each data collection period (baseline, follow up at month 2, follow up at month 4). Sedentary and MVPA cut points for children will be used to measure of the mean amplitude deviation of acceleration [Vaha-Ypya 2015].
Change in parent-child feeding practices | Baseline (pre-intervention), Month 2 (post-intervention), Month 4 (follow up)
  The Food Parenting Inventory (FPI) [Power et al 2019] measures food parenting practices and has been validated among diverse populations. We will utilize 5 subscales that link specifically to our HEROs curriculum including: Encourages Exploration of New Foods (3 items), Offers New Foods (3 items), Repeatedly Presents New Foods (3 items), Pressure to Eat (4 items) and Food as Reward (3 items). Response options are a 5-point Likert scale (never to always). The mean score per FPI scale will be calculated for analyses.
Change in physical activity parenting practices | Baseline (pre-intervention), Month 2 (post-intervention), Month 4 (follow up)
  The Preschooler's Physical Activity Parenting Practices (PPAPP) instrument [O'Connor et al 2014] has been validated in a large sample of parents of preschoolers. The Engagement/Structure sub-scale (15 items), and 2 single-items (Have outdoor toys; Not enrolled in sports-reverse coded) measures parenting practices that encourage child physical activity. Practices that discourage child physical activity include 4 subscales: Promote Inactivity (3 items), Promote Screen Time (3 items), Psychological Control (5 items), and Restriction for Safety Concerns (4 items). Response options are a 5-point Likert scale (never to always). A mean score per PPAPP scale will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Laura L Bellows, PhD, Principal Investigator — Colorado State University; Susan L Johnson, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Colorado State University, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: Undecided
Data may be available upon request to the Principal Investigator

REFERENCES:
- [Background] Vaha-Ypya H, Vasankari T, Husu P, Manttari A, Vuorimaa T, Suni J, Sievanen H. Validation of Cut-Points for Evaluating the Intensity of Physical Activity with Accelerometry-Based Mean Amplitude Deviation (MAD). PLoS One. 2015 Aug 20;10(8):e0134813. doi: 10.1371/journal.pone.0134813. eCollection 2015. PMID 26292225
- [Background] Power TG, Johnson SL, Beck AD, Martinez AD, Hughes SO. The Food Parenting Inventory: Factor structure, reliability, and validity in a low-income, Latina sample. Appetite. 2019 Mar 1;134:111-119. doi: 10.1016/j.appet.2018.11.033. Epub 2018 Nov 30. PMID 30508613
- [Background] Johnson SL, Ryan SM, Kroehl M, Moding KJ, Boles RE, Bellows LL. A longitudinal intervention to improve young children's liking and consumption of new foods: findings from the Colorado LEAP study. Int J Behav Nutr Phys Act. 2019 Jun 3;16(1):49. doi: 10.1186/s12966-019-0808-3. PMID 31159810
- [Background] Townsend MS, Shilts MK, Styne DM, Drake C, Lanoue L, Ontai L. An Obesity Risk Assessment Tool for Young Children: Validity With BMI and Nutrient Values. J Nutr Educ Behav. 2018 Jul-Aug;50(7):705-717. doi: 10.1016/j.jneb.2018.01.022. Epub 2018 Mar 19. PMID 29567008
- [Background] O'Connor TM, Cerin E, Hughes SO, Robles J, Thompson DI, Mendoza JA, Baranowski T, Lee RE. Psychometrics of the preschooler physical activity parenting practices instrument among a Latino sample. Int J Behav Nutr Phys Act. 2014 Jan 15;11:3. doi: 10.1186/1479-5868-11-3. PMID 24428935
- [Background] Logan SW, Robinson LE, Getchell N. The comparison of performances of preschool children on two motor assessments. Percept Mot Skills. 2011 Dec;113(3):715-23. doi: 10.2466/03.06.25.PMS.113.6.715-723. PMID 22403917